CLINICAL TRIAL: NCT00461981
Title: A Phase 2, Prospective, Randomized, Open-Label Study to Evaluate the Immune Responses of FluMist® Compared With Trivalent Inactivated Vaccine (TIV) in Children 12 to <36 Months of Age
Brief Title: A Phase 2 Study to Evaluate Immune Responses of FluMist®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Maria Allende, M.D., MedImmune Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP128
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2010-01

CONDITIONS: Influenza Vaccine
Keywords: Live, attenuated influenza virus vaccine (LAIV); Trivalent inactivated influenza virus vaccine (TIV); FluMist
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FluMist, Influenza Virus Vaccine Live (Experimental): FluMist, Influenza Virus Vaccine Live, Intranasal
  Interventions: Biological: FluMist, Influenza Virus Vaccine Live
- TIV, Trivalent Inactivated Influenza Virus Vaccine (Active Comparator): TIV, Trivalent Inactivated Influenza Virus Vaccine, Intramuscular
  Interventions: Biological: TIV, Trivalent Inactivated Influenza Virus Vaccine

INTERVENTIONS:
Biological: TIV, Trivalent Inactivated Influenza Virus Vaccine — 0.25 mL will be administered intramuscularly for each of two doses
  Arms: TIV, Trivalent Inactivated Influenza Virus Vaccine
Biological: FluMist, Influenza Virus Vaccine Live — 0.5 mL will be administered intranasally (approximately 0.25 mL into each nostril) for each of two doses
  Arms: FluMist, Influenza Virus Vaccine Live

SUMMARY:
The primary objective of this study is to describe the level of serum antibody and cellular immune responses conferred by FluMist and TIV against influenza virus strains.

DETAILED DESCRIPTION:
The primary objective of this study is to describe the level of serum antibody and cellular immune responses conferred by FluMist and TIV against antigenically matched and antigenically mismatched influenza virus strains.

The secondary objective of this study is to describe the safety of FluMist and TIV in subjects 12 to <36 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 12 to <36 months (reached their 1st year but not yet reached their 3rd year birthday) at the time of randomization
* Written informed consent and HIPAA authorization obtained from the subject's legal representative
* Ability of the subject's legal representative to understand and comply with the requirements of the study
* Subject's legal representative available by telephone
* Ability to complete follow-up period of 180 days after final study vaccination as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of FluMist or TIV, including egg or egg products
* History of hypersensitivity to gentamicin
* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy
* Household contact who is immunocompromised (participants should also avoid close contact with immunocompromised individuals for at least 21 days after each study vaccination)
* History of Guillain-Barré syndrome
* Any prior history of wheezing or asthma
* Acute febrile (≥100.0°F oral or equivalent) and/or clinically significant respiratory illness (e.g., cough or sore throat) within 72 hours prior to either study vaccination
* Use of aspirin or aspirin-containing products within the 30 days prior to randomization, or expected receipt through 180 days after final study vaccination
* Receipt of any prior influenza vaccine
* Use of anti-influenza medications (including amantadine, rimantadine, oseltamivir, and zanamivir) within 14 days prior to randomization, or expected receipt through 35 days after final study vaccination
* Administration of any live virus vaccine, other than measles, mumps, rubella, and varicella-containing vaccine(s), within 30 days prior to randomization, or expected receipt through 30 days after final study vaccination
* Administration of any inactivated (i.e., non-live) vaccine within 14 days prior to randomization, or expected receipt within 14 days before or 14 days after either study vaccination
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 180 days after final study vaccination (use of licensed agents for indications not listed in the package insert is permitted)
* Receipt of any blood product within 90 days prior to randomization, or expected receipt through 35 days after final study vaccination
* Family member or household contact who is an employee of the research center or otherwise involved with the conduct of the study
* Any condition that in the opinion of the investigator would interfere with evaluation of the vaccine or interpretation of study results

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Allende, M.D., Study Director — MedImmune LLC
Locations (19):
- United States (19):
  - Harvey Pediatrics, Jonesboro, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - NuLife Clinical Research, Anaheim, California
  - Palm Beach Research Center, West Palm Beach, Florida
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Peak Medical Research, LLC, Owensboro, Kentucky
  - Benchmark Research, Metairie, Louisiana
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Henderson Pediatrics, Henderson, Nevada
  - Regional Clinical Research, Inc., Endwell, New York
  - Dayton Clinical Research, Dayton, Ohio
  - Northeast Cincinnati Pediatric Asso., Inc., Mason, Ohio
  - Celia Reyes-Acuna, M.D., Corpus Christi, Texas
  - Allergy Immunology Research Center of North Texas, Dallas, Texas
  - Healthcare Discoveries, Inc., San Antonio, Texas
  - Wee Care Pediatrics, Layton, Utah
  - Bear Care Pediatrics, Ogden, Utah
  - Advanced Pediatrics, Vienna, Virginia
  - Pediatrics at the Beach, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 101 subjects were entered and randomized into the study at 15 sites in the United States of America between 07 May 2007 and 28 Jun 2007.
Groups:
- FluMist, Influenza Virus Vaccine Live: FluMist, Influenza Virus Vaccine Live, Intranasal, 0.25 mL will be administered intranasally for each of two doses
- TIV, Trivalent Inactivated Influenza Virus Vaccine: TIV, Trivalent Inactivated Influenza Virus Vaccine, Intramuscular, 0.25 mL will be administered intramuscularly for each of two doses
Period: Overall Study
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Started | 50 | 51
Completed | 39 | 42
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 9 | 6
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: months] | 23.1 (7.0) | 24.4 (7.0) | 23.8 (7.0)
Age, Customized [Number; unit: participants]
  12 to < 24 months | 26 | 24 | 50
  24 to < 36 months | 24 | 27 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 28 | 30 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 16 | 38
  White | 26 | 31 | 57
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 44 | 42 | 86
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI)Seroconversion Following the First Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days post Dose 1 (n=44; n=40), no major protocol violations (n=44; n=39), and had a baseline HAI titer of 4 or less (n=24; n=27).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 24 | 27
Percentage of Participants | 20.8 | 81.5
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; The seroconversion rates (the proportions of baseline seronegative subjects achieving a 4 or more fold increase in titer from baseline) were summarized for baseline seronegative subjects by treatment group and by dose number. A two-sided exact 95% confidence interval (CI) was constructed on the rate differences using the unconditional exact method proposed by Chan and Zhang (Chan, 1999); Test type: Superiority or Other; Rate differences = -60.6, 95% CI [-79.7 to -31.7]

2. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the Second Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=23; n=26), no major protocol violations (n=23; n=26), and had a baseline HAI titer of 4 or less (n=14; n=19).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 14 | 19
Percentage of Participants | 28.6 | 89.5
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = -60.9, 95% CI [-83.8 to -26.0]

3. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI)Seroconversion Following the First Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /ca A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days post Dose 1 (n=44; n=40), no major protocol violations (n=42; n=39), and had a baseline HAI titer of 4 or less (n=20; n=26).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 20 | 26
Percentage of Participants | 75.0 | 30.8
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = 44.2, 95% CI [12.0 to 67.8]

4. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI)Seroconversion Following the Second Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /ca A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=23; n=26), no major protocol violations (n=21; n=26), and had a baseline HAI titer of 4 or less (n=13; n=19).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 13 | 19
Percentage of Participants | 84.6 | 68.4
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = 16.2, 95% CI [-17.6 to 45.4]

5. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI)Seroconversion Following the First Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Wisconsin/67/05 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days post Dose 1 (n=44; n=40), no major protocol violations (n=43; n=40), and had a baseline HAI titer of 4 or less (n=34; n=30).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 34 | 30
Percentage of Participants | 61.8 | 80.0
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = -18.2, 95% CI [-40.0 to 4.9]

6. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the Second Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Wisconsin/67/05 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=23; n=26), no major protocol violations (n=22; n=26), and had a baseline HAI titer of 4 or less (n=18; n=18).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 18 | 18
Percentage of Participants | 94.4 | 100
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = -5.6, 95% CI [-27.4 to 13.3]

7. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the First Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the B /wt B/Malaysia/2506/04 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days post Dose 1 (n=44; n=40), no major protocol violations (n=44; n=37), and had a baseline HAI titer of 4 or less (n=34; n=31).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 34 | 31
Percentage of Participants | 64.7 | 29.0
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = 35.7, 95% CI [9.5 to 57.1]

8. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the Second Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the B /wt B/Malaysia/2506/04 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=23; n=26), no major protocol violations (n=23; n=25), and had a baseline HAI titer of 4 or less (n=20; n=20).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 90.0 | 95.0
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = -5.0, 95% CI [-27.7 to 16.0]

9. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the First Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/Solomon Island/3/06 antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days post Dose 1 (n=44; n=40), no major protocol violations (n=43; n=39), and had a baseline HAI titer of 4 or less (n=24; n=29).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 24 | 29
Percentage of Participants | 25.0 | 10.3
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = 14.7, 95% CI [-6.5 to 38.4]

10. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the Second Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /wt A/Solomon Island/3/06 antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=23; n=26), no major protocol violations (n=22; n=26), and had a baseline HAI titer of 4 or less (n=14; n=21).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 14 | 21
Percentage of Participants | 71.4 | 33.3
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = 38.1, 95% CI [0.9 to 65.9]

11. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the First Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Brisbane/10/2007 antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days post Dose 1 (n=44; n=40), no major protocol violations (n=43; n=40), and had a baseline HAI titer of 4 or less (n=36; n=31).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 36 | 31
Percentage of Participants | 47.2 | 35.5
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = 11.7, 95% CI [-13.0 to 34.9]

12. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Hemagglutination Inhibition (HAI) Seroconversion Following the Second Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Brisbane/10/2007 antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=23; n=26), no major protocol violations (n=22; n=26), and had a baseline HAI titer of 4 or less (n=19; n=19).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 19 | 19
Percentage of Participants | 78.9 | 94.7
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = -15.8, 95% CI [-40.7 to 8.0]

13. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 24 | 27
Titer | 4.4 [2.59 to 8.23] | 10.1 [7.60 to 13.37]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; Corresponding two-sided 95% CIs based on 10,000 bootstrap data sets for the ratios of strain-specific GMTs (FluMist/TIV) were constructed by drawing replicates with replacement from each of the 2 cells (2 treatment groups) of observed data. The number of replicates drawn from each cell in this fashion was equal to the observed sample size within each cell. For each of the 10,000 bootstrap data sets, the overall GMT ratio was calculated; Test type: Superiority or Other; GMT ratio = 0.43, 95% CI [0.24 to 0.87]

14. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2)for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 14 | 19
Titer | 6.2 [3.12 to 13.13] | 30.9 [19.92 to 46.09]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.20, 95% CI [0.09 to 0.48]

15. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /ca A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 20 | 26
Titer | 19.0 [10.56 to 34.30] | 5.7 [3.69 to 9.39]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMT Ratio = 3.36, 95% CI [1.54 to 7.13]

16. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /ca A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 13 | 19
Titer | 37.6 [19.80 to 67.51] | 11.5 [6.91 to 19.20]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT ratio = 3.26, 95% CI [1.44 to 7.19]

17. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Wisconsin/67/05 Influenza Strain antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 34 | 30
Titer | 12.5 [7.53 to 21.28] | 11.8 [8.38 to 17.15]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 1.06, 95% CI [0.56 to 1.96]

18. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Wisconsin/67/05 Influenza Strain antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 18 | 18
Titer | 27.4 [16.63 to 43.55] | 47.0 [30.79 to 69.12]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.58, 95% CI [0.31 to 1.12]

19. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the B /wt B/Malaysia/2506/04 Influenza Strain antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 34 | 31
Titer | 9.8 [6.52 to 15.36] | 4.1 [3.20 to 5.35]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 2.40, 95% CI [1.48 to 3.97]

20. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the B /wt B/Malaysia/2506/04 Influenza Strain antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 20 | 20
Titer | 16.0 [10.56 to 24.25] | 33.1 [21.86 to 50.21]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.48, 95% CI [0.27 to 0.87]

21. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/Solomon Island/3/06 Influenza Strain antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 24 | 29
Titer | 4.2 [2.75 to 7.23] | 2.9 [2.15 to 4.30]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 1.45, 95% CI [0.80 to 2.66]

22. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /wt A/Solomon Island/3/06 Influenza Strain antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 14 | 21
Titer | 8.0 [4.42 to 14.49] | 4.6 [3.17 to 6.78]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 1.75, 95% CI [0.88 to 3.39]

23. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Brisbane/10/2007 Influenza Strain antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 36 | 31
Titer | 7.0 [4.49 to 11.10] | 4.7 [3.27 to 7.00]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 1.49, 95% CI [0.80 to 2.69]

24. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The HAI GMTs of baseline seronegative subjects (baseline titer of 4 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Brisbane/10/2007 Influenza Strain antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 19 | 19
Titer | 10.7 [6.91 to 16.59] | 17.2 [11.11 to 26.66]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.62, 95% CI [0.33 to 1.16]

25. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the First Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days after Dose 1 (n=41; n=40), no major protocol violations (n=40; n=34), and had a baseline HAI titer of 10 or less (n=19; n=18).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 19 | 18
Percentage of Participants | 26.3 | 72.2
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate differences = -45.9, 95% CI [-71.7 to -11.6]

26. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the Second Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=22; n=26), no major protocol violations (n=21; n=19), and had a baseline HAI titer of 10 or less (n=12; n=12).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 12 | 12
Percentage of Participants | 75.0 | 100
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = -25.0, 95% CI [-57.2 to 4.8]

27. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the First Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /ca A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days after Dose 1 (n=41; n=40), no major protocol violations (n=40; n=35), and had a baseline HAI titer of 10 or less (n=20; n=20).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 80.0 | 15.0
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = 65.0, 95% CI [34.4 to 85.3]

28. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the Second Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /ca A/New Caledonia/20/999 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=22; n=26), no major protocol violations (n=20; n=22), and had a baseline HAI titer of 10 or less (n=12; n=13).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 12 | 13
Percentage of Participants | 91.7 | 92.3
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = -0.6, 95% CI [-30.4 to 30.3]

29. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the First Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Wisconsin/67/05 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days after Dose 1 (n=41; n=40), no major protocol violations (n=35; n=31), and had a baseline HAI titer of 10 or less (n=27; n=21).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 27 | 21
Percentage of Participants | 63.0 | 100
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = -37.0, 95% CI [-57.8 to -17.5]

30. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the Second Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Wisconsin/67/05 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=22; n=26), no major protocol violations (n=17; n=22), and had a baseline HAI titer of 10 or less (n=12; n=16).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 12 | 16
Percentage of Participants | 91.7 | 100
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = -8.3, 95% CI [-38.5 to 14.5]

31. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the First Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the B /wt B/Malaysia/2506/04 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days after Dose 1 (n=41; n=40), no major protocol violations (n=30; n=27), and had a baseline HAI titer of 10 or less (n=22; n=21).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 22 | 21
Percentage of Participants | 40.9 | 19.0
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = 21.9, 95% CI [-6.7 to 48.1]

32. Primary Outcome: Percentage of Subjects With Antigenically Matched Strain-specific Microneutralization Seroconversion Following the Second Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the B /wt B/Malaysia/2506/049 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=22; n=26), no major protocol violations (n=16; n=16), and had a baseline HAI titer of 10 or less (n=13; n=12).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 13 | 12
Percentage of Participants | 69.2 | 91.7
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = -22.4, 95% CI [-54.4 to 12.2]

33. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Microneutralization Seroconversion Following the First Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/Solomon Island/3/06 antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days after Dose 1 (n=41; n=40), no major protocol violations (n=16; n=14), and had a baseline HAI titer of 10 or less (n=1; n=3).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 1 | 3
Percentage of Participants | 100 | 66.7
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = 33.3, 95% CI [-81.1 to 90.6]

34. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Microneutralization Seroconversion Following the Second Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /wt A/Solomon Island/3/06 antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=22; n=26), no major protocol violations (n=7; n=8), and had a baseline HAI titer of 10 or less (n=1; n=2).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 1 | 2
Percentage of Participants | 100 | 100
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = 0.0, 95% CI [-97.5 to 84.2]

35. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Microneutralization Seroconversion Following the First Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Brisbane/10/2007 antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-42 days after Dose 1 (n=41; n=40), no major protocol violations (n=7; n=12), and had a baseline HAI titer of 10 or less (n=3; n=7).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 3 | 7
Percentage of Participants | 33.3 | 42.9
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = -9.5, 95% CI [-65.2 to 58.8]

36. Primary Outcome: Percentage of Subjects With Antigenically Mismatched Strain-specific Microneutralization Seroconversion Following the Second Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The percentage of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Brisbane/10/2007 antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: The immunogenicity (IM) population included all subjects who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had valid IM assay results obtained at baseline and at 28-35 days post Dose 2 (n=22; n=26), no major protocol violations (n=7; n=8), and had a baseline HAI titer of 10 or less (n=5; n=5).
Measure: Number; unit: Percentage of Participants
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 5 | 5
Percentage of Participants | 80.0 | 100
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Rate difference = -20.0, 95% CI [-71.6 to 33.9]

37. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 19 | 18
Titer | 10.7 [8.47 to 13.60] | 47.5 [32.90 to 67.24]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.23, 95% CI [0.15 to 0.35]

38. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H1N1 /wt A/New Caledonia/20/99 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /wt A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 12 | 12
Titer | 24.5 [15.87 to 37.75] | 226.2 [126.95 to 391.60]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.11, 95% CI [0.05 to 0.22]

39. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /ca A/New Caledonia/20/99 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 20 | 20
Titer | 56.6 [31.39 to 101.96] | 11.7 [9.16 to 15.68]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 4.85, 95% CI [2.51 to 9.22]

40. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H1N1 /ca A/New Caledonia/20/99 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /ca A/New Caledonia/20/999 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 12 | 13
Titer | 164.4 [79.63 to 339.03] | 49.6 [33.30 to 68.39]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 3.31, 95% CI [1.46 to 7.54]

41. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Wisconsin/67/05 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 27 | 21
Titer | 83.1 [37.46 to 177.29] | 61.4 [45.64 to 82.68]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 1.35, 95% CI [0.58 to 3.04]

42. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H3N2 /wt A/Wisconsin/67/05 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Wisconsin/67/05 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 30
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 12 | 16
Titer | 190.1 [75.41 to 415.10] | 433.3 [287.10 to 653.93]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.44, 95% CI [0.16 to 1.07]

43. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the B /wt B/Malaysia/2506/04 antigenically matched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 22 | 21
Titer | 21.9 [12.24 to 41.82] | 8.9 [6.72 to 12.39]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 2.46, 95% CI [1.26 to 5.06]

44. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H1N1 /wt A/Solomon Island/3/06 antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 1 | 3
Titer | 28.0 [28.00 to 28.00] | 31.5 [28.00 to 40.00]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.89, 95% CI [0.70 to 1.00]

45. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - B /wt B/Malaysia/2506/04 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the B /wt B/Malaysia/2506/049 antigenically matched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 13 | 12
Titer | 34.0 [18.39 to 71.81] | 67.1 [42.12 to 105.14]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.51, 95% CI [0.23 to 1.22]

46. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H1N1 /wt A/Solomon Island/3/06 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H1N1 /wt A/Solomon Island/3/06 antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 34
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 1 | 2
Titer | 160.0 [160.00 to 160.00] | 40.0 [40.00 to 40.00]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 4.00, 95% CI [4.00 to 4.00]

47. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the First Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 1 (28-42 days after Dose 1) for the H3N2 /wt A/Brisbane/10/2007 antigenically mismatched influenza strain
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: as for outcome 35
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 3 | 7
Titer | 22.4 [10.00 to 113.00] | 28.2 [15.50 to 56.59]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.80, 95% CI [0.22 to 3.63]

48. Primary Outcome: Microneutralization Geometric Mean Titers (GMTs) in Baseline Seronegative Subjects Following the Second Dose - H3N2 /wt A/Brisbane/10/2007 Influenza Strain
Description: The microneutralization GMTs of baseline seronegative subjects (baseline titer of 10 or less) achieving a 4 or more fold increase in titer from baseline at Post Dose 2 (28-35 days after Dose 2) for the H3N2 /wt A/Brisbane/10/2007 antigenically mismatched influenza strain
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: as for outcome 36
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 5 | 5
Titer | 56.3 [24.38 to 121.20] | 85.8 [52.85 to 129.87]
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.66, 95% CI [0.25 to 1.73]

49. Primary Outcome: Immunogenicity Response by B-cell IgG and IgA ELISPOT Assay
Description: Counts of antibody secreting cells (ASCs) per 10^6 peripheral blood mononuclear cells (PBMCs) for influenza-specific response (ie, anti-IgG fluorescein [FLU] or anti-IgA FLU) and influenza-specific response after adjusting plate background response (ie, anti-IgG FLU/anti-IgG total or anti-IgA FLU/anti-IgA total) as measured by B-cell ELISPOT assay at 7 to 10 days after Dose 1
Time Frame: Post Dose 1 (7 to 10 days post Dose 1)
Population: Evaluable subjects for the ELISPOT immunogenicity included those who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had baseline data (n=30; n=35), and any protocol-specified post-dose timepoint data for B-cell ELISPOT (n=16; n=17).
Measure: Median (Full Range); unit: Counts of ASCs per 10^6 PBMCs
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 16 | 17
Counts of ASCs per 10^6 PBMCs
  Anti-IgG FLU | 6.5 [0.0 to 574.5] | 57.0 [0.0 to 556.5]
  Anti-IgG FLU/Anti-IgG Total | 0.030 [0.000 to 0.796] | 0.204 [0.000 to 2.200]
  Anti-IgA FLU | 4.8 [0.0 to 49.5] | 22.0 [0.0 to 82.0]
  Anti-IgA FLU/Anti-IgA Total | 0.011 [0.000 to 0.161] | 0.043 [0.000 to 0.300]

50. Primary Outcome: Immunogenicity Response by B-cell IgG and IgA ELISPOT Assay
Description: Counts of antibody secreting cells (ASCs) per 10^6 peripheral blood mononuclear cells (PBMCs) for influenza-specific response (ie, anti-IgG fluorescein [FLU] or anti-IgA FLU) and influenza-specific response after adjusting plate background response (ie, anti-IgG FLU/anti-IgG total or anti-IgA FLU/anti-IgA total) as measured by B-cell ELISPOT assay at 7 to 10 days after Dose 2
Time Frame: Post Dose 2 (7 to 10 days post Dose 2)
Population: Evaluable subjects for the ELISPOT immunogenicity included those who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV), had baseline data (n=30; n=35), and any protocol-specified post-dose timepoint data for B-cell ELISPOT (n=10; n=9).
Measure: Median (Full Range); unit: Counts of ASCs per 10^6 PBMCs
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 10 | 9
Counts of ASCs per 10^6 PBMCs
  Anti-IgG FLU | 45.5 [13.0 to 212.0] | 45.0 [0.0 to 350.0]
  Anti-IgG FLU/Anti-IgG Total | 0.161 [0.017 to 0.530] | 0.076 [0.000 to 2.000]
  Anti-IgA FLU | 7.0 [0.0 to 53.0] | 7.0 [0.0 to 33.0]
  Anti-IgA FLU/Anti-IgA Total | 0.015 [0.003 to 0.094] | 0.018 [0.000 to 0.075]

51. Primary Outcome: Median Fold-Rises in the Number of Interferon-gamma Elispots Per 200,000 Peripheral Blood Mononuclear Cells (PBMCs) by T-cell Elispot Assay Following the First Dose
Description: Median number of PBMCs secreting interferon-gamma as measured by the number of spot forming cells per 200,000 PBMCs (SPC/2 x 10^5 PBMCs) as measured by the T-cell Elispot assay at 28 to 42 days after Dose 1. The results were summarized for wild-type (wt) influenza-specific response (wt fluorescein [FLU]) after adjusting plate background response at 28 to 42 days after Dose 1
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Population: Evaluable subjects for the ELISPOT immunogenicity included those who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV) and had valid pre-Dose 1 and post-Dose 1 T-cell Elispot results (n=12; n=15)
Measure: Median (Full Range); unit: SPC/2 x 10^5 PBMCs
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 12 | 15
SPC/2 x 10^5 PBMCs | 3.3 [0.3 to 6.0] | 1.2 [0.1 to 155.1]

52. Primary Outcome: Median Fold-Rises in the Number of Interferon-gamma Elispots Per 200,000 Peripheral Blood Mononuclear Cells (PBMCs) by T-cell Elispot Assay
Description: Median number of PBMCs secreting interferon-gamma as measured by the number of spot forming cells per 200,000 PBMCs (SPC/2 x 10^5 PBMCs) as measured by the T-cell Elispot assay at 28 to 35 days after Dose 2. The results were summarized for wild-type (wt) influenza-specific response (wt fluorescein [FLU]) after adjusting plate background response at 28 to 35 days after Dose 2
Time Frame: Post Dose 2 (28 to 35 days post Dose 2)
Population: Evaluable subjects for the ELISPOT immunogenicity included those who received at least 1 full dose of study vaccine (n=50 for FluMist; n=51 for TIV) and had valid pre-Dose 1 and any post-Dose T-cell Elispot results (n=3; n=6)
Measure: Median (Full Range); unit: SPC/2 x 10^5 PBMCs
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 3 | 6
SPC/2 x 10^5 PBMCs | 3.6 [0.8 to 4.8] | 3.2 [2.2 to 14.6]

53. Primary Outcome: Distribution of Interferon (IFN)-Alpha/Beta Gene Signature Scores Among All Subjects
Description: Distribution of IFN-alpha/beta gene signature scores at 7 to 10 days after Dose 1. IFN alpha/beta gene signature scores were calculated as the average fold change in a panel of 21 type 1 IFN-inducible genes. The distribution of IFN alpha/beta gene signature scores ranged from -4 to 4, with -4 representing the lowest level of activity and 4 representing the highest level of activity. The percentage of subjects by IFN-alpha/beta gene signature score for each treatment group were compared.
Time Frame: Post Dose 1 (28 to 42 days post Dose 1)
Measure: Number; unit: Units on a scale
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Number analyzed (Participants) | 43 | 42
Units on a scale
  Gene signature score of -4 (%) | 0.02 | 0.00
  Gene signature score of -3 (%) | 0.00 | 0.00
  Gene signature score of -2 (%) | 0.02 | 0.02
  Gene signature score of -1 (%) | 0.07 | 0.29
  Gene signature score of 0 (%) | 0.23 | 0.57
  Gene signature score of 1 (%) | 0.21 | 0.07
  Gene signature score of 2 (%) | 0.21 | 0.05
  Gene signature score of 3 (%) | 0.14 | 0.00
  Gene signature score of 4 (%) | 0.09 | 0.00
Statistical Analysis 1: Comparison: FluMist, Influenza Virus Vaccine Live vs TIV, Trivalent Inactivated Influenza Virus Vaccine; Test type: Non-Inferiority or Equivalence — Equivalence; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of administration of the first dose of study vaccine (Study Day 0) through 42 days after administration of the final dose.
Description: Legal representatives were given worksheets to capture AEs. The study staff contacted the subject's legal representative at the scheduled clinic visits and 28 to 35 days post Dose 2 to collect AEs. A telephone contact occurred at 43 to 57 days after administration of the final dose of study vaccine to collect AEs through 42 days.
Arm/Group | FluMist, Influenza Virus Vaccine Live | TIV, Trivalent Inactivated Influenza Virus Vaccine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 26/50 | 31/51
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FluMist, Influenza Virus Vaccine Live (N=50) | TIV, Trivalent Inactivated Influenza Virus Vaccine (N=51)
Arthropod Bite (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Irritability (General disorders) | 2 (2) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 11 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (12)
Teething (Gastrointestinal disorders) | 1 (1) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.